CLINICAL TRIAL: NCT04966364
Title: Investigation of the Effect of Applying Hypotension Prediction Index Guidance for Prevention of Intraoperative Hypotension During Major Gastrointestinal Surgery: A Randomized Trial
Brief Title: Hypotension Prediction Index in Major Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 202105065RINA
Record Dates: First submitted 2021-07-14; First posted 2021-07-19 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2021-07

CONDITIONS: the Effect of Hypotension Prediction Index Application

STUDY DESIGN:
Intervention Model Description: using hypotension prediction index guided in the operation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participants and care provider and outcome assessor are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with hypotension prediction index guided (Active Comparator): Patients receiving hypotension prediction index guided. In this group, they will be alerted when the index exceeded 85 (range 0 to 100) indicating the later occurrence of MAP< 65mmHg for at least minutes and a treatment protocol based on advanced hemodynamic parameters recommended vasopressor or inotrope, fluid administration, or observation.
  Interventions: Device: hypotension prediction index guided
- patients without hypotension prediction index gudied (Other): Patients will receive usual care during the operation without hypotension prediction index alerted.
  Interventions: Device: without hypotesion prediction index guided

INTERVENTIONS:
Device: hypotension prediction index guided — patients receiving hypotension prediction index monitoring and let the anesthesiologist' alerted the coming intraoperatiobe hypotension
  Arms: patients with hypotension prediction index guided
Device: without hypotesion prediction index guided — patients receiving usual care without hypotension prediction index monitoring but with usual arterial line care
  Arms: patients without hypotension prediction index gudied

SUMMARY:
Intraoperative hypotension (IOH) is defined as a mean arterial pressure (MAP) of < 65mmHg during surgery. Patients undergoing major gastrointestinal (GI) surgery, such as esophagectomy with reconstruction, are at a high-risk of IOH because such surgeries typically require more than 3h to complete and require blood transfusion or inotrope administration. Critically, these surgeries involve organ removal or substitute connection, which require wound or flap anastomosis. IOH is believed to be associated with postoperative anastomosis necrosis. It increases the risk of postoperative intrathoracic or abdominal infection, resulting in septic shock, postoperative major organ dysfunction and mortality.

The data of TWA-MAP< 65mmHg in the HPI guidance group will be significantly lower than that in the group without HPI guidance.

DETAILED DESCRIPTION:
Intraoperative hypotension (IOH) is defined as a mean arterial pressure (MAP) of < 65mmHg during surgery. Patients undergoing major gastrointestinal (GI) surgery, such as esophagectomy with reconstruction, are at a high-risk of IOH because such surgeries typically require more than 3h to complete and require blood transfusion or inotrope administration. Critically, these surgeries involve organ removal or substitute connection, which require wound or flap anastomosis. IOH is believed to be associated with postoperative anastomosis necrosis. It increases the risk of postoperative intrathoracic or abdominal infection, resulting in septic shock, postoperative major organ dysfunction and mortality.

The Hypotension Prediction Index (HPI) is an algorithm made commercially available in 2019. On the basis of arterial waveform features, HPI predicts hypotension defined as MAP < 65 mmHg for at least 1 min. In two previous randomized trials(RCTs), the primary outcome was the severity and duration of hypotension, defined as a time-weighted average mean arterial pressure (TWA-MAP) less than 65 mmHg (formula: (total area under MAP<65mmHg(mmHg*hours))/(surgery length (hours));normal range:0.01-0.5mmHg).A higher data of TWA-MAP<65mmHg indicates severe and longer IOH. However, according to the results of the previous two RCTs, the effects of HPI guidance during surgery remain inconclusive.

We aim to investigate whether HPI guidance can be used to reduce the duration and severity of hypotension during major GI surgery. Our hypothesis is that the data of TWA-MAP< 65mmHg in the HPI guidance group will be significantly lower than that in the group without HPI guidance. Postoperative major complications and mortality will be followed.

Methods: Sixty patients aged 20 to 80 years undergoing elective GI surgery will be randomized to receive hemodynamic management with or without HPI guidance. Clinicians caring for patients assigned to the HPI guidance group will be alerted when the index exceeded 85 (range 0 to 100) indicating the later occurrence of MAP< 65mmHg for at least minutes and a treatment protocol based on advanced hemodynamic parameters recommended vasopressor or inotrope, fluid administration, or observation. Primary outcome is the data of TWA-MAP<65mmHg. Postoperative complications will be recorded on postoperative day 3,7 and 30. The mortality rate from the time of hospitalization to postoperative 30 days will be recorded.

The data of TWA-MAP< 65mmHg in the HPI guidance group will be significantly lower than that in the group without HPI guidance.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving elective major gastrointestinal surgery

Exclusion Criteria:

* emergent surgery
* pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
time-weighted average mean arterial pressure less than 65 mmHg | during the operation
  .A higher data of time-weighted average mean arterial pressure less than 65 mmHg indicates severe and longer intraoperative hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No
due to the ethical concern

REFERENCES:
- [Derived] Lai CJ, Cheng YJ, Han YY, Hsiao PN, Lin PL, Chiu CT, Lee JM, Tien YW, Chien KL. Hypotension prediction index for prevention of intraoperative hypotension in patients undergoing general anesthesia: a randomized controlled trial. Perioper Med (Lond). 2024 Jun 15;13(1):57. doi: 10.1186/s13741-024-00414-7. PMID 38879506